CLINICAL TRIAL: NCT03326583
Title: The Effects of Patiromer on Serum Potassium Level and Gut Microbiome of End Stage Renal Disease Patients With Hyperkalemia
Brief Title: The Effects of Patiromer on Serum Potassium Level and Gut Microbiome of ESRD Patients With Hyperkalemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dominic Raj (Other)
Responsible Party: Sponsor-Investigator, Dominic Raj, Director of the Division of Renal Disease and Hypertension, Professor of Medicine, George Washington University
Organization: George Washington University (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 071738
Record Dates: First submitted 2017-10-06; First posted 2017-10-31 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-04

CONDITIONS: ESRD; Hyperkalemia; End Stage Renal Disease
Keywords: End Stage Renal Disease; ESRD; Hyperkalemia
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperkalemia | interventions — patiromer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patiromer (Experimental): This arm is a 2 week observation period before the start of the Patiromer treatment phase, followed by a 12 week treatment phase, and 6 week no treatment observation phase.
  Pre-Treatment (Wk 1-2): Observational period. Baseline sample collection of blood and stool. No medication.
  Treatment (Wk 3-14): Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks. Blood and stool will be collected.
  Post-Treatment (Wk 15-20): Observational period. No medication. Blood and stool will be collected.
  Interventions: Drug: Patiromer

INTERVENTIONS:
Drug: Patiromer — Patiromer will be orally self-administered by participants.

SUMMARY:
The Effects of Patiromer on Serum Potassium Level and Gut Microbiome of ESRD Patients With Hyperkalemia (potassium greater than 5 milliequivalents per liter) is a non-randomized, crossover study. This is an open-label, pilot clinical trial with 3 sequential phases of (a) 2 weeks of no intervention, (b) 12 weeks of Patiromer treatment, and (c) 6 weeks of no intervention. Treatment with Patiromer will be initiated at a dose of 8.4 grams, once daily and observed for a week, then uptitrated to 16.8 grams once daily. Eligible study subjects will collect stool samples and provide blood and urine samples.

ELIGIBILITY:
Inclusion Criteria:

* Subjects on stable hemodialysis for more than 90 days.
* Age 18-85 years.
* Persistent hyperkalemia, defined as elevated serum potassium > 5.0 mEq/L in more than 2 occasions during the previous 3 months.

Exclusion Criteria:

* Use of pre- or probiotics during the past 2 months
* Use of antibiotics within the past 2 months, if the patient received a single course of antibiotic.
* Presence of chronic wound infection and osteomyelitis
* Inflammatory bowel disease, chronic diarrhea, current C. difficile infection
* Liver cirrhosis or chronic active hepatitis
* Treatment with immunosuppressive medications in the past 6 months or more than a week of treatment with prednisone > 10 mg in the last 3 months
* Anticipated kidney transplant within 9 months
* Expected survival < 9 months
* Pregnancy, anticipated pregnancy, or breastfeeding
* Incarceration
* Participation in another intervention study
* severe anemia defined as hemoglobin < 8.0 g/dl any time during the last 2 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- DaVita K Street, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Amdur RL, Paul R, Barrows ED, Kincaid D, Muralidharan J, Nobakht E, Centron-Vinales P, Siddiqi M, Patel SS, Raj DS. The potassium regulator patiromer affects serum and stool electrolytes in patients receiving hemodialysis. Kidney Int. 2020 Nov;98(5):1331-1340. doi: 10.1016/j.kint.2020.06.042. Epub 2020 Aug 1. PMID 32750456

RESULTS

PARTICIPANT FLOW:
Groups:
- Patiromer: This arm is the 2 week observation period before the start of the Patiromer treatment phase, followed by a 12 week treatment phase, and 6 week no treatment observation phase.
  Pre-Treatment (Wk 1-2): Observational period. Baseline sample collection of blood and stool. No medication.
  Treatment (Wk 3-14): Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks. Blood and stool will be collected.
  Post-Treatment (Wk 15-20): Observational period. No medication. Blood and stool will be collected.
  Patiromer: Patiromer will be orally self-administered by participants.
Period: Pre-Treatment
Arm/Group | Patiromer
Started | 27
Completed | 26
Not Completed | 1
Period: Treatment
Arm/Group | Patiromer
Started | 26
Completed | 24
Not Completed | 2
Period: Post-Treatment
Arm/Group | Patiromer
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patiromer
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33 (7)
Diabetes [Count of Participants; unit: Participants] | 11
Coronary Artery Disease [Count of Participants; unit: Participants] | 3
HIV [Count of Participants; unit: Participants] | 5
Heart Failure [Count of Participants; unit: Participants] | 2
Hemoglobin [Mean (Standard Deviation); unit: g/dl] | 10.8 (1.3)
Mean Corpuscular Volume (MCV) [Mean (Standard Deviation); unit: femtoliters] | 90.8 (9.7)
Whole Blood Count (WBC) [Mean (Standard Deviation); unit: 1000 cells/microliters] | 6.4 (1.8)
Blood Urea Nitrogen [Mean (Standard Deviation); unit: mg/dl] | 60.9 (15.9)
Creatinine [Mean (Standard Deviation); unit: mg/dl] | 10.2 (2)
Sodium [Mean (Standard Deviation); unit: mEq/L] | 138.4 (3.1)
Potassium [Mean (Standard Deviation); unit: mEq/L] | 5.6 (.6)
Bicarbonate [Mean (Standard Deviation); unit: mEq/L] | 20.2 (2.9)
Calcium [Mean (Standard Deviation); unit: mg/dL] | 8.9 (.7)
Phosphate [Mean (Standard Deviation); unit: mg/dL] | 6.0 (1.8)
Glucose [Mean (Standard Deviation); unit: mg/dL] | 120.7 (59.6)
Parathyroid hormone (PTH) [Mean (Standard Deviation); unit: pg/ml] | 333.7 (254.6)
Magnesium [Mean (Standard Deviation); unit: mg/dL] | 2.6 (.5)
Total Protein [Mean (Standard Deviation); unit: g/dL] | 7.1 (.6)
Serum Albumin [Mean (Standard Deviation); unit: g/dL] | 4.1 (.2)
Kt/V [Mean (Standard Deviation); unit: ratio] | 1.4 (.2)
Dialysate potassium [Mean (Standard Deviation); unit: mEq/L] | 2.0 (.2)
Dialysate sodium [Mean (Standard Deviation); unit: mEq/L] | 136.2 (.9)
Dialysate calcium [Mean (Standard Deviation); unit: mEq/dL] | 2.5 (.1)
Erythropoietin dose [Mean (Standard Deviation); unit: UI/mL] — units 3 times weekly
  UI/mL | 6200 (2699)
Dialysate magnesium [Mean (Standard Deviation); unit: mEq/L] | 1 (0)
Doxercalciferol [Mean (Standard Deviation); unit: micrograms] — 3 times weekly
  micrograms | 3.6 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events of Participants Taking Patiromer in Lowering Serum Potassium Levels in End Stage Renal Disease (ESRD) Patients With Hyperkalemia Measured by Gastrointestinal Symptom Rating Scale (GSRS)
Description: The Gastrointestinal Symptom Rating Scale was used to measures any potential side effects due to study medication. Survey was administered at Wk 1, Wk 8, Wk 14, and Wk 20.
  For symptoms (abdomen pain - diarrhea) a score of 0 indicates "no discomfort", 1 = "mild discomfort", 2=moderate, 3=severe; higher score means a worse outcome
  For stool form, 1=Well formed, 2=Semi formed, 3= Loose, 4= Liquid;higher score means a worse outcome
  For number of stools per day, 1= <1, 2=1 or 2, 3=3 or 4, 4=5 or 6,5= 7 or more; higher score means a worse outcome
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-Treatment)
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Pre-Treatment: 2 week observation period before treatment
- Treatment: 12 week treatment phase, . Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks.
  Patiromer: Patiromer will be orally self-administered by participants.
- Post-Treatment: 6 week follow up, off medication
Arm/Group | Pre-Treatment | Treatment | Post-Treatment
Number analyzed (Participants) | 27 | 24 | 24
score on a scale
  Abdomen Pain | .24 [.04 to .44] | .23 [0 to .51] | .16 [0 to .32]
  Heartburn | .08 [0 to .17] | .31 [.02 to .59] | .13 [0 to .32]
  Acid Reflux | .22 [.03 to .41] | .35 [.06 to .64] | .30 [.04 to .56]
  Hunger Pains | 0 [0 to 0] | .19 [0 to .38] | .04 [0 to .13]
  Nausea | .44 [.14 to .75] | .42 [.11 to .74] | .14 [0 to .39]
  Rumbling Stomach | .34 [.14 to .54] | .23 [0 to .48] | .31 [0 to .62]
  Bloated | .14 [0 to .28] | .12 [0 to .24] | .14 [0 to .28]
  Burping | .13 [.02 to .25] | .08 [0 to .18] | .26 [0 to .57]
  Flatus | .53 [.18 to .88] | .58 [.21 to .94] | .60 [.18 to 1.02]
  Constipation | .72 [.31 to 1.12] | .65 [.23 to 1.08] | .36 [0 to .72]
  Diarrhea | .17 [.03 to .32] | .44 [.06 to .82] | .18 [.02 to .34]
  Stool form | 1.43 [1.20 to 1.66] | 1.62 [1.39 to 1.84] | 1.41 [1.14 to 1.68]
  Number of stool/days | 1.9 [1.7 to 2.2] | 2.1 [1.8 to 2.4] | 2 [1.8 to 2.2]
Statistical Analysis 1: Comparison: Pre-Treatment vs Treatment vs Post-Treatment; Test type: Superiority; p = .05, Fisher Exact

2. Primary Outcome: Serum Potassium Level Through 12 Weeks of Treatment
Description: Blood was collected during Pre-Treatment week 2, Treatment Week 14, and Post-Treatment week 20
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-Treatment)
Measure: Mean (95% Confidence Interval); unit: mEq/L
Groups:
- Pre-Treatment: 2 week observational period before starting medication
- Intervention: Treatment: Treatment (Wk 14): Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks. Blood and stool will be collected.
- Post-Treatment: Wk 20 (6 weeks off treatment)
  Post-Treatment (Wk 20): Observational period. No medication. Blood and stool will be collected.
Arm/Group | Pre-Treatment | Intervention: Treatment | Post-Treatment
Number analyzed (Participants) | 27 | 24 | 24
mEq/L | 5.7 [5.4 to 5.9] | 5.1 [4.9 to 5.2] | 5.4 [5.2 to 5.6]
Statistical Analysis 1: Comparison: Pre-Treatment vs Intervention: Treatment vs Post-Treatment; Test type: Superiority; p = .05, Mixed Models Analysis

3. Primary Outcome: Changes in Blood Chemistry During the Study
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-Treatment)
Measure: Mean (95% Confidence Interval); unit: mg/dl
Groups:
- Treatment: Week 14 (12 weeks of treatment), . Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks.
  Patiromer: Patiromer will be orally self-administered by participants.
- Post-Treatment: Wk 20 (6 week follow up off medication)
Arm/Group | Pre-Treatment | Treatment | Post-Treatment
Number analyzed (Participants) | 27 | 24 | 24
mg/dl
  Blood Urea Nitrogen | 62.2 [56.9 to 67.5] | 62.6 [57.3 to 67.9] | 59.0 [54.1 to 64.0]
  Creatinine | 10.4 [9.7 to 11.0] | 10.6 [9.9 to 11.4] | 10.5 [9.9 to 11.1]
  Sodium | 138.4 [137.3 to 139.5] | 138.5 [137.5 to 139.6] | 139.2 [135.7 to 142.6]
  Potassium | 5.7 [5.4 to 5.9] | 5.1 [4.9 to 5.2] | 5.4 [5.2 to 5.6]
  Chloride | 95.2 [94.0 to 96.5] | 95.1 [94.0 to 96.3] | 95.8 [94.6 to 97.0]
  Carbon Dioxide | 20.3 [19.4 to 21.2] | 20.0 [19.1 to 20.9] | 20.6 [19.5 to 21.7]
  Calcium | 8.9 [8.7 to 9.1] | 9.1 [8.9 to 9.4] | 8.7 [8.5 to 8.9]
  Phosphate | 6.0 [5.3 to 6.7] | 6.0 [5.4 to 6.7] | 6.3 [5.7 to 7.0]
  Magnesium | 2.6 [2.4 to 2.8] | 2.4 [2.3 to 2.6] | 2.5 [2.4 to 2.7]
Statistical Analysis 1: Comparison: Pre-Treatment vs Treatment vs Post-Treatment; Test type: Superiority; p = .05, Mixed Models Analysis

4. Primary Outcome: Stool Electrolytes During the Study Phases
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-Treatment)
Measure: Mean (95% Confidence Interval); unit: mcg/g
Groups:
- Treatment: Treatment (Wk 14): Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks. Blood and stool will be collected.
Arm/Group | Pre-Treatment | Treatment | Post-Treatment
Number analyzed (Participants) | 27 | 24 | 24
mcg/g
  Sodium | 343 [222 to 464] | 425 [288 to 562] | 360 [241 to 479]
  Potassium | 4132 [3627 to 4637] | 5923 [4796 to 7050] | 4246 [3858 to 4634]
  Calcium | 7874 [5799 to 9948] | 13017 [10448 to 15586] | 7635 [5568 to 9703]
  Phosphate | 7719 [6630 to 8809] | 7067 [5780 to 8354] | 7670 [6341 to 8998]
  Magnesium | 1923 [1380 to 2466] | 1603 [1347 to 1860] | 1665 [1372 to 1958]
Statistical Analysis 1: Comparison: Pre-Treatment vs Treatment vs Post-Treatment; Test type: Superiority; p = .05, Mixed Models Analysis

5. Secondary Outcome: Changes in Plasma Metabolites Using p-Cresol of Hyperkalemic ESRD Patients Treated With Patiromer
Description: Blood and stool samples collected from the ESRD patient will be collected at pre-specified time points and analyzed by untargeted and targeted metabolomics for stool and serum metabolome profiles.
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-Treatment)
Population: Targeted metabolomic analysis using p-cresol were not performed due to financial constraints.
Arm/Group | Pre-Treatment | Treatment | Post-Treatment
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Changes in Gut Microbiome of Hyperkalemic ESRD Patients Treated With Patiromer.
Description: Blood and stool samples collected from the ESRD patient will be collected at pre-specified time points and analyzed by metagenomics for gut microbiome profile.
Time Frame: Wk 2 (Pre-Treatment), Wk 14 (Treatment), Wk 20 (Post-treatment)
Population: Targeted metabolomic analyses using p-cresol were not performed due to financial constraints.
Arm/Group | Pre-Treatment | Treatment | Post-Treatment
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The study period during which adverse events must be reported is defined as the period from initiation of the study procedures to the end of the treatment follow-up. In other words, AE documentation should begin when the patient signs the informed consent form. Encourage participants to contact the investigator after the conclusion of the trial if subsequent medical events occur which the participant, or the participant's physician, believes may be related to participation in the research study
Description: The center staff will collect adverse event data at each study visit by checking several different sources of information by asking participants directly, evaluating medical record information, reviewing all laboratory values, examining reports generated by the data management system based on data entered into logs and forms.
  AE information may also be reported between scheduled study visits via regular contacts if the participant reports health related problems or concerns
Groups:
- Patiromer: This arm is the 2 week observation period before the start of the Patiromer treatment phase, followed by a 12 week treatment phase, and 6 week no treatment observation phase.
  Pre-Treatment (Wk 1-2): Observational period. Baseline sample collection of blood and stool. No medication.
  Treatment (Wk 3-14): Participants will take 8.4 grams of Patiromer once daily for one week, during which serum potassium and gastrointestinal symptoms will be evaluated. If tolerated and in the absence of hypokalemia, the dose will be up-titrated to 16.8 grams once daily for the remaining 11 weeks. Blood and stool will be collected.
  Post-Treatment (Wk 15-20): Observational period. No medication. Blood and stool will be collected.
Arm/Group | Patiromer
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 11/27
Other Adverse Events (participants affected / at risk) | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=27)
Hypoglycemia (Metabolism and nutrition disorders) | 1 — Pt was admitted to the hospital Sunday, 11/19/17 after collapsing at a relatives house. He was diagnosed with hypoglycemia. Potassium was 5.9. Pt began study drug on 11/15/17 but did not take in hospital. Pt also had high glucose, 400. Pt doing well
Hypertension (Cardiac disorders) | 1 — Pt send to the emergency department mid dialysis with hypertensive urgency and headache. Given 20 mg IV hydralazine, which decreased BP. Pt was discharged on 2/14.
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 — Pt presented in ED with SOB and cough, has history of asthma and seasonal allergies. Treated with steroids and albuterol. Drug not taking during hospitalization.
Fever (Infections and infestations) | 1 — Pt presented in Ed post dialysis with 6 days of fever, headache, sore throat, R side neck pain. Blood test revealed methicillin-resistant staphylococcus aureus (MRSA ) infection. Ppt treated with antibiotics
Hypoglcymia (Metabolism and nutrition disorders) | 1 — Pt arrived at dialysis feeling drowsy, blood sugar was 41, admitted to ED where treated with glucose and food. Glucose levels improved and patient returned to normal dialysis.
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 — Patient admitted to the hospital for shortness of breath and hyperkalemia (8.0). Pt treated with Veltessa.
MRSA Infection (Infections and infestations) | 1 — Pt reported being hospitalized during the week of July 27, 2018 for MRSA. Pt reported being treated with antibiotics.
Infection (Infections and infestations) | 1 — Pt admitted to hospital for arteriovenous (AV) fistula infection. Pt discharged on 10/10/18. Pt was off medication from 10/3-10/5.
Dizzy and Disoriented (General disorders) | 1 — Pt had been complaining of feeling dizzy and disoriented w/o nausea. Bloodwork and MRI came back normal. Pt treated for vertigo and discharged.
Nasuea (Gastrointestinal disorders) | 1 — Pt presented to ER on 11/14/19 with nausea/vomiting and shortness of breath (SOB). No findings on imagining studies. Pt dx w/ intractable vomiting w/ mild epigastric tenderness. Treated with ondansetron and metoclopramide and discharged
Right Arm Collulitis (Skin and subcutaneous tissue disorders) | 1 — Pt presented to ER@ request of dialysis unit. Pt c/o R arm swelling, pain, erythema. Treated with vancomycin and compression wrap. Discharged with antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patiromer (N=27)
hypomagnesemia (Metabolism and nutrition disorders) | 0
constipation (Gastrointestinal disorders) | 0
diarrhea (Gastrointestinal disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-25): https://cdn.clinicaltrials.gov/large-docs/83/NCT03326583/Prot_SAP_000.pdf